CLINICAL TRIAL: NCT02028559
Title: Safety and Effectiveness of the Ultrasonic Propulsion of Kidney Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jonathan Harper, MD, Assistant Professor, Urology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00002746
Record Dates: First submitted 2014-01-01; First posted 2014-01-07 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Kidney Stones; Nephrolithiasis; Urolithiasis
Keywords: stones; kidney; stone fragments; lithotripsy
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Urolithiasis; Calculi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessors a) evaluating imaging for stone growth, b) evaluating relatedness of safety events to the device/procedure or underlying stone condition, and c) evaluating relapse events are blind to the exposure condition.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment with Ultrasonic Propulsion (Experimental): Subjects receive treatment with the Propulse 1 device. Intervention consists of the non-invasive application of ultrasound to move stones within the kidney and ureter.
  Interventions: Device: Propulse 1
- Control (No Intervention): Subject follow same protocol as treatment group but do not receive the ultrasonic propulsion intervention.

INTERVENTIONS:
Device: Propulse 1 — Move kidney stones with Propulse 1 device.
  Arms: Treatment with Ultrasonic Propulsion

SUMMARY:
This study tests moving kidney stones using focused ultrasound (referred to as ultrasonic propulsion). The study includes multiple population groups to investigate the ability of our technology to: a) move stone fragments to a location within the kidney to improve their chances of passage, and thus reduce the occurrence of additional symptomatic events and retreatment or b) move a symptomatic stone to relieve symptoms and pain.

DETAILED DESCRIPTION:
This is an investigator initiated, NIH-funded study conducted by the University of Washington (UW). Our research group has developed a new, non-invasive technology using low intensity focused ultrasound to reposition kidney stones by imparting sufficient acoustic energy to physically move a stone. The focused ultrasound pulses are similar to pulses that may be used in elastography or acoustic radiation force imaging. Like conventional ultrasound, the probe is placed in contact with the patient's skin to image the stone following standard ultrasound imaging procedure. The same probe is then used to focus the ultrasound and apply a burst (a sequence of pulses) of acoustic force to push the stone. Brightness mode (B-mode) imaging is interleaved with the "pushing" pulses (Push-mode) to monitor stone movement. The user controls the burst amplitude. To limit heating at the probe surface, there is a slight delay before the operator can execute the next push.

In addition to undergoing the investigational procedure, the research activities include the following:

* subjects undergo a pain questionnaire before and after the procedure;
* the subject's skin in the area of probe placement is observed before and after the procedure;
* subjects are contacted once-a-week for 3 weeks to evaluate for potential adverse events, pain medication use, and, if applicable, stone passage;
* subjects are requested to undergo at least one follow-up imaging 4 - 12 weeks post-procedure;
* a review of each subject's medical records is conducted 90-days post-procedure to evaluate for additional effectiveness and safety events.
* Specifically for the residual fragment population (randomized control trial), subjects are contacted every 6 months for 3 years and their charted is reviewed for 5 years for stone growth, symptomatic, unscheduled medical visits, and surgery related to stones.

Subjects that qualify for the trial are recruited into different study arms (referred to as Population groups) based on their type of stone condition (de novo stone versus post-lithotripsy fragment), size of stone (≤ 5 mm or > 5 mm), and management plan (clinical observation or surgical intervention). The objectives vary based upon the Population group. Subjects may qualify for more than one population group over time and may undergo the investigational procedure up to 4 times total (inclusive of both the left and right-side urinary tracts). Population groups 1-3 has been closed. Therefore, the details provided for this registration is for Population group 4.

1. First-in-Human Population (Closed): This was the initial group of subjects included under this clinical trial. This was a 15-subject feasibility that included a broad range of populations. This feasibility population formulated the basis for expanding the trial into a larger study addressing each population separately. This is encompassed in subject populations 2-5 below.
2. Acute Subject Population (Closed): All subjects undergo the investigational procedure. Subjects undergo the investigational procedure awake and in the clinic or emergency department (ED) setting. To qualify the subject must have clinical imaging confirmation of an obstructing stone with their pain managed and complete a urinalysis to assess infection risk. Ultrasonic propulsion is used with the intent to relieve the obstruction and associated pain. A subset of subjects were exposed to higher amplitude dislodging pulses, in addition to the ultrasonic propulsion pulses.
3. De Novo Subject Population (Closed): Subjects undergo the investigational procedure awake and in the clinic. To qualify the subject must have a de novo stone ≤ 5 mm or, if larger, be scheduled for surgical intervention on the same day. Ultrasonic propulsion is used with the intent to help facilitate stone passage (≤ 5 mm) or demonstrate the ability to move larger stones. In the case of subjects scheduled for URS, the investigative procedure can be conducted concurrently with the standard-of-care procedure (see bullet point #2 above).
4. URS Subject Population (Closed): Subjects undergo the investigational procedure while anesthetized and concurrently undergoing a ureteroscopy guided laser lithotripsy procedure (referred to herein as URS). To qualify the subject must have at least one stone ≤ 20 mm in the largest dimension and be scheduled for surgery. Ultrasonic propulsion may be used to move a de novo stone or stone fragments of varying sizes generated over the course of the URS procedure. Note that since these subjects are anesthetized, a pain questionnaire is not included as part of their protocol.
5. Residual Fragment Population: Subjects undergo the investigational procedure awake and in the clinic setting. To qualify the subject must have at least one residual fragment (≤ 5 mm in largest dimension) identified either on imaging or based on the investigator's interpretation of that imaging. This is a prospective, open-label, multicenter, randomized control trial (RCT) with a treatment arm and control arm. The only difference in protocol between the two arms is that only the treatment group undergoes the investigational procedure and the associated post-procedure pain questionnaire and the post-procedure skin surface inspection. Ultrasonic propulsion is used with the intent to demonstrate the ability of the ultrasonic propulsion device to reposition stones within the human kidney and the subsequent clinical benefit of facilitating stone passage and reducing stone burden to reduce relapse. This is the only population group recruited across more than one site - the UW and the VA Puget Sound Heathcare System.

The final data set collected from the study will be analyzed under two separate statistical analysis plan (SAPs) referred to as NIH SAP and Pivotal SAP.

ELIGIBILITY:
Inclusion Criteria:

* Individuals suspected of having at least one stone remaining from the lithotripsy procedure
* Individuals at least 4-weeks post-lithotripsy procedure
* Individuals with residual stone fragments ≤ 5 mm in largest dimension (individually)
* Individuals being managed with watchful waiting or medical therapy for stones

Primary Exclusion Criteria:

* Individuals under 18 years of age
* Individuals with non-echogenic stones
* Individuals unable or unwilling to comply with the follow-up requirements
* Individuals with a coagulation abnormality or taking blood thinners or other anticoagulant at clinically significant levels
* Individuals with mobility issues who are unable to comfortably lie for up to 30 minutes or roll from their back to their side
* Individuals belonging to a vulnerable group (pregnant, mentally disabled, physically disabled, prisoner, etc.)
* Individuals who have already received four previous ultrasonic propulsion procedures.
* Individuals who have received an ultrasonic propulsion treatment within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of relapse | Measurement over 3-year follow-up (phone call or email encounter semi-annually) and 5-year review of the subject's medical records, including imaging (no subject participation).
  The primary outcome measure (NIH SAP) is the proportion of subjects experiencing relapse defined as: an unscheduled, symptomatic visit for stones on the study side, future surgery for stones on the study side, or stone growth of a residual fragment measured by clinical imaging exams.
Measurement of stone passage | Measurement occurs over 3 weeks (weekly phone call or email encounter with the subject) plus review of the subject's medical chart).
  The primary effectiveness outcome measure (Pivotal SAP) is the proportion of subjects reporting visual observation of stone passage during the 3-week follow-up period after initial treatment (Treatment Group) or randomization (Control Group).
Measurement of low frequency adverse events of interest | Measurement over 3 weeks (weekly phone call or email encounter with the subject) plus review of the subject's medical chart).
  The primary safety outcome measure (Pivotal SAP) is subject-level rate of low frequency adverse events (AEs) of interest defined as skin burn, clinically significant hematuria, renal injury requiring intervention, clinically significant hematoma, sepsis, or any other procedure or device related event meeting the definition of a serious adverse event (SAE) with onset after the initial procedure (Treatment Group) or randomization (Control Group).

SECONDARY OUTCOMES:
Measurement of all adverse effects associated with the procedure | Measurement over 3 weeks (weekly phone call or email encounter with the subject) plus review of the subject's medical chart.
  The study measures the subject-level rate of adverse events with onset after the procedure (Treatment group) or randomization (Control group) through the 3-week follow-up determined by a blinded reviewer to be potentially related to the device, procedure, or the subject's underlying kidney disease. (Secondary endpoint for both SAPs).

OTHER OUTCOMES:
Measurement of stone motion caused by ultrasound | At the time of treatment. To be evaluated with each treatment pulse over an approximately 1-hour study.
  The study will measure the extent of stone motion from the real-time ultrasound images. This information will be used to establish any relationships between stone motion and stone passage.
Measurement of discomfort related to the procedure | At the time of treatment. To be evaluated over an approximately 1 hour study.
  The subject will be asked directly what feeling or discomfort, if any, they experienced with each the treatment pulses. The subject will be asked to fill out a pain questionnaire before and after the research study.
Measurement of the reduction in stone burden based on imaging | Measurement occurs at baseline through study completion, which is up to 5 years.
  The study will measure any decrease in stone burden based on post-procedure (Treatment group) or post-randomization (Control group) imaging to establish any relationship between stone passage and a change in stone burden on imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Harper, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - VA Puget Sound Health Care System, Seattle, Washington
  - University of Washington Department of Urology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hall MK, Thiel J, Dunmire B, Samson PC, Kessler R, Sunaryo P, Sweet RM, Metzler IS, Chang HC, Gunn M, Dighe M, Anderson L, Popchoi C, Managuli R, Cunitz BW, Burke BH, Ding L, Gutierrez B, Liu Z, Sorensen MD, Wessells H, Bailey MR, Harper JD. First Series Using Ultrasonic Propulsion and Burst Wave Lithotripsy to Treat Ureteral Stones. J Urol. 2022 Nov;208(5):1075-1082. doi: 10.1097/JU.0000000000002864. Epub 2022 Nov 1. PMID 36205340
- [Result] Dai JC, Sorensen MD, Chang HC, Samson PC, Dunmire B, Cunitz BW, Thiel J, Liu Z, Bailey MR, Harper JD. Quantitative Assessment of Effectiveness of Ultrasonic Propulsion of Kidney Stones. J Endourol. 2019 Oct;33(10):850-857. doi: 10.1089/end.2019.0340. Epub 2019 Sep 25. PMID 31333058
- [Result] Harper JD, Cunitz BW, Dunmire B, Lee FC, Sorensen MD, Hsi RS, Thiel J, Wessells H, Lingeman JE, Bailey MR. First in Human Clinical Trial of Ultrasonic Propulsion of Kidney Stones. J Urol. 2016 Apr;195(4 Pt 1):956-64. doi: 10.1016/j.juro.2015.10.131. Epub 2015 Oct 30. PMID 26521719
- [Derived] Sorensen MD, Dunmire B, Thiel J, Cunitz BW, Burke BH, Levchak BJ, Popchoi C, Holmes AE, Kucewicz JC, Hall MK, Dighe M, Dai JC, Cormack FC, Liu Z, Bailey MR, Porter MP, Harper JD. Randomized Controlled Trial of Ultrasonic Propulsion-Facilitated Clearance of Residual Kidney Stone Fragments vs Observation. J Urol. 2024 Dec;212(6):811-820. doi: 10.1097/JU.0000000000004186. Epub 2024 Aug 15. PMID 39146526
- [Derived] Harper JD, Metzler I, Hall MK, Chen TT, Maxwell AD, Cunitz BW, Dunmire B, Thiel J, Williams JC, Bailey MR, Sorensen MD. First In-Human Burst Wave Lithotripsy for Kidney Stone Comminution: Initial Two Case Studies. J Endourol. 2021 Apr;35(4):506-511. doi: 10.1089/end.2020.0725. Epub 2020 Nov 5. PMID 32940089
- See also: Related Info — http://apl.uw.edu/pushingstones